CLINICAL TRIAL: NCT05781750
Title: A Phase 2b, Randomized, Controlled Double-blind, Multicenter Study Comparing the Efficacy and Safety of Zetomipzomib (KZR-616) 30 mg or 60 mg With Placebo in Patients With Active Lupus Nephritis
Brief Title: A Study of Zetomipzomib (KZR-616) in Patients With Active Lupus Nephritis (PALIZADE)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision.
Sponsor: Kezar Life Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KZR-616-202
Record Dates: First submitted 2023-03-12; First posted 2023-03-23 (Actual); Results first posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Lupus Nephritis
Keywords: immunoproteasome inhibition; selective immunoproteasome inhibition; complete renal response; partial renal response; glucocorticoids; steroids; SLE (systemic lupus erythematosus); UPCR (urine protein to creatinine ratio); eGFR (estimated glomerular filtration rate)
MeSH Terms: conditions — Lupus Nephritis; Lupus Erythematosus, Systemic | interventions — KZR-616

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- zetomipzomib 30 mg + standard-of-care (Experimental): Participants randomized to be treated with initial 30 mg dose of zetomipzomib, followed by weekly doses of 30 mg zetomipzomib through the treatment period in addition to background standard of care therapy.
  Interventions: Drug: zetomipzomib
- zetomipzomib 60 mg + standard-of-care (Experimental): Participants randomized to be treated with initial 30 mg dose of zetomipzomib, followed by weekly doses of 60 mg zetomipzomib through the treatment period in addition to background standard of care therapy.
  Interventions: Drug: zetomipzomib
- placebo + standard-of-care (Placebo Comparator): Participants randomized to be treated with initial 30 mg dose of placebo, followed by weekly doses (30 mg or 60 mg) of placebo through the treatment period in addition to background standard of care therapy.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: zetomipzomib — Subcutaneous injection of zetomipzomib
  Other Names: KZR-616
  Arms: zetomipzomib 30 mg + standard-of-care; zetomipzomib 60 mg + standard-of-care
Drug: placebo — Subcutaneous injection of placebo
  Other Names: matching placebo
  Arms: placebo + standard-of-care

SUMMARY:
The purpose of this study was to assess the efficacy and safety of zetomipzomib (30 mg or 60 mg) compared with placebo in achieving renal response after 52 weeks of treatment in patients with active lupus nephritis (LN).

DETAILED DESCRIPTION:
This study aimed to investigate whether zetomipzomib, added to standard of care treatment in patients with active LN, was able to reduce disease activity over a treatment period of 52 weeks. The background standard of care therapy was mycophenolate mofetil (MMF) and initial optional treatment with IV methylprednisolone, followed by a tapering course of oral corticosteroids.

Patients were required to have a diagnosis of LN according to established diagnostic criteria and clinical and biopsy features suggestive of active nephritis.

Patients were randomized in a 2:1 ratio to receive either zetomipzomib (30 mg or 60 mg) or placebo administered as a subcutaneous injection once weekly for 52 weeks, followed by a 4-week safety follow-up period. Efficacy was to be assessed by measuring the level of proteinuria (as measured by urine protein to creatinine ratio [UPCR]) and estimated glomerular filtration rate (eGFR) as compared to current standard of care treatment. Safety was also assessed throughout the study to ensure an acceptable safety profile.

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index of ≥18 kg/m^2
* eGFR ≥30 mL/min/1.73 m^2
* Unequivocally positive ANA test result and/or a positive anti-dsDNA serum antibody test
* Diagnosis of LN according to 2003 or 2018 ISN/RPS criteria and confirmed by renal biopsy performed within 12 months prior to Screening.
* UPCR ≥1.0 (Class III/IV +/-V) or UPCR ≥2.0 (Class V)
* Adequate hematologic, hepatic, and renal function

Key Exclusion Criteria:

* Current or medical history of:

  * Central nervous system manifestations of SLE
  * Overlapping autoimmune condition that may affect study assessments/outcomes
  * Antiphospholipid syndrome with history of thromboembolic event of within the 52 weeks prior to Screening
  * Thrombocytopenia or at high risk for developing clinically significant bleeding or organ dysfunction requiring therapies (i.e., plasmapheresis or acute blood or platelet transfusions
  * Solid organ transplant or planned transplant during study
  * Malignancy of any type, with exceptions for non-melanoma skin cancers and certain cancers >5 years ago
* Has received dialysis within the 52 weeks prior to Screening
* Positive test at Screening for HIV, hepatitis B/C
* Known intolerance to MMF or equivalent and corticosteroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2023-11-03 (Actual); Primary Completion 2024-11-08 (Actual); Study Completion 2024-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kezar, Study Director — Kezar Life Sciences, Inc.
Locations (49):
- United States (4):
  - Accurate Clinical Research - Lake Charles, Lake Charles, Louisiana
  - Nephrology Associates, Inc, East Providence, Rhode Island
  - Precision Comprehensive Clinical Research Solutions, Colleyville, Texas
  - Prolato Clinical Research Center (PCRC), Houston, Texas
- Argentina (7):
  - Mayo Clinic of UCMB SRL, San Miguel de Tucumán, Tucumán Province
  - Framingham Medical Center, Buenos Aires
  - Medical Research Organization, Buenos Aires
  - Aprillus Assistance and Research by Arcis Health, Buenos Aires
  - Dr. Doreski Medical Offices, Buenos Aires
  - Military Central Hospital, Buenos Aires
  - Austral University Hospital, Pilar
- Brazil (4):
  - Holy House of Mercy of Belo Horizonte, Belo Horizonte, Minas Gerais
  - Clinics Hospital FMRP, Ribeirão Preto, São Paulo
  - Faculty of Medicine of SJRP, São José do Rio Preto, São Paulo
  - Clinical Hospital FMUSP, São Paulo
- China (3):
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
- Costa Clinica, Barranquilla, Atlántico, Colombia
- Laiko General Hospital of Athens, Athens, Greece
- Guatemala (3):
  - Center for Advanced Health Clinical Studies, Guatemala City
  - Clinical Research Center, S.A., Guatemala City
  - Medical Clinic Specialized in Internal Medicine and Rheumatology, Guatemala City
- India (13):
  - All India Institute of Medical Sciences, Raipur, Chhattisgarh
  - Nirmal Hospital, Surat, Guajrat
  - Unity Hospital, Surat, Guajrat
  - Panchshil Hospital, Ahmedabad, Gujarat
  - Elite Mission Hospital, Thrissur, Kerala
  - MGM Medical College and Hospital, Aurangabad, Maharashtra
  - Kingsway Hospital, Nagpur, Maharashtra
  - Jasleen Hospital, Nagpur, Maharashtra
  - Assured Care Plus Hospital, Nashik, Maharashtra
  - Sir Ganga Ram Hospital, New Delhi, NCT of Delhi
  - SMS Medical College, Jaipur, Rajasthan
  - Yashoda Hospitals, Hyderabad, Telangana
  - Krishna Institute of Medical Science, Secunderabad, Telangana
- Malaysia (5):
  - Prince Court Medical Centre, Kuala Lumpur, Kuala Lumpur
  - Hospital Raja Permaisuri Bainun, Ipoh, Perak
  - Hospital Selayang, Batu Caves, Selangor
  - Hospital Sultan Idris Shah Serdang, Kajang, Selangor
  - University Malaya Medical Centre, Kuala Lumpur
- Philippines (6):
  - Mary Mediatrix Medical Center, Lipa City, Batangas
  - Iloilo Doctors' Hospital, Iloilo City, Iloilo
  - ManilaMed - Medical Center Manila, Manila, National Capital Region
  - St. Luke's Medical Center, Quezon City, National Capital Region
  - Far Eastern University Hospital Nicanor Reyes Medical Foundation, Quezon City, National Capital Region
  - University of Santo Tomas Hospital, Manila
- Phoenix Pharma, Port Elizabeth, Eastern Cape, South Africa
- The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Corporate website — https://www.kezarlifesciences.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Zetomipzomib 30 mg + Standard-of-care | Zetomipzomib 60 mg + Standard-of-care | Placebo + Standard-of-care
Started | 27 | 29 | 28
Completed | 0 | 0 | 0
Not Completed | 27 | 29 | 28

BASELINE CHARACTERISTICS:
Population: Among the 11 participants who were stratified to Pure Class V LN, one was actually diagnosed as Class IV and was mistakenly stratified to Pure Class V. All primary and secondary outcome measures are presented as stratified, whereas the post-hoc outcome measures include the participant who was stratified incorrectly.
Groups:
- Total: Total of all reporting groups
Arm/Group | Zetomipzomib 30 mg + Standard-of-care | Zetomipzomib 60 mg + Standard-of-care | Placebo + Standard-of-care | Total
Number analyzed (Participants) | 27 | 29 | 28 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.0 (10.54) | 32.5 (9.44) | 32.8 (9.10) | 32.1 (9.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 28 | 25 | 78
  Male | 2 | 1 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 10 | 13 | 28
  Not Hispanic or Latino | 22 | 19 | 15 | 56
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 5 | 2 | 8
  Asian | 19 | 15 | 13 | 47
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 3 | 5
  White | 6 | 7 | 9 | 22
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 2
Average 24-hour UPCR at Screening [Count of Participants; unit: Participants]
  ≤3.0 mg/mg | 13 | 15 | 13 | 41
  >3.0 mg/mg | 14 | 14 | 15 | 43
Average 24-hour UPCR at Baseline [Mean (Standard Deviation); unit: mg/mg] | 3.7 (2.0) | 3.6 (2.1) | 3.1 (1.6) | 3.5 (1.9)
SLEDAI-2K [Mean (Standard Deviation); unit: score on a scale] — Scale from 0-105, higher scores indicate worse disease.
  score on a scale | 11.8 (5.28) | 11.7 (5.48) | 10.5 (5.02) | 11.3 (5.23)
Time from SLE diagnosis to Screening [Mean (Standard Deviation); unit: years] | 4.7 (5.0) | 8.1 (6.2) | 6.7 (5.8) | 6.5 (5.8)
Time from LN diagnosis to Screening [Mean (Standard Deviation); unit: years] | 1.8 (2.3) | 5.0 (5.4) | 4.3 (4.5) | 3.7 (4.5)
LN Class [Number; unit: participants]
  Class III/IV ± V | 23 | 26 | 24 | 73
  Pure Class V | 4 | 3 | 4 | 11

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Achieving Complete Renal Response
Description: Proportion of patients achieving complete renal response (CRR), defined as:
  * A UPCR ≤0.5 in one 24-hour urine sample (for primary endpoint and Week 53) or 2 consecutive first morning void urine samples (for all other time points)
  * An eGFR ≥60 mL/min/1.73 m^2 or no confirmed decrease of >20% from Baseline eGFR.
Time Frame: Week 37
Population: Participants in the intent to treat analysis set who reached Week 37 of treatment. Intent-to-treat set was defined as the set of all participants who are randomized to the study. This analysis focuses on the participants with Class III/IV ± Class V lupus nephritis. Due to the early termination of the study, not all participants reached the 37 week timepoint for efficacy analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Zetomipzomib 30 mg + Standard-of-care | Zetomipzomib 60 mg + Standard-of-care | Placebo + Standard-of-care
Number analyzed (Participants) | 4 | 6 | 6
Participants | 0 | 1 | 0

2. Secondary Outcome: Proportion of Patients Achieving Partial Renal Response (PRR)
Description: Proportion of patients achieving PRR, defined as a:
  ≥50% reduction of UPCR from Baseline, and to <1.0 if the Baseline UPCR was <3.0 or to <3.0 if the Baseline value was ≥3.0.
Time Frame: Week 25 and Week 37
Population: Participants in the intent to treat set, defined as the set of all participants who are randomized to the study. This analysis focuses on the participants with Class III/IV ± Class V lupus nephritis. Due to the early termination of the study, not all participants reached the timepoints for efficacy analysis and no participants completed the full 52-week treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | Zetomipzomib 30 mg + Standard-of-care | Zetomipzomib 60 mg + Standard-of-care | Placebo + Standard-of-care
Number analyzed (Participants) | 16 | 15 | 15
Participants
  Week 25 | 5 | 8 | 6
  Week 37: number analyzed (Participants) | 4 | 6 | 6
  Week 37 | 1 | 1 | 0

3. Secondary Outcome: Proportion of Patients Achieving Complete Renal Response
Description: Proportion of patients achieving complete renal response (CRR)
Time Frame: Week 25
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Zetomipzomib 30 mg + Standard-of-care | Zetomipzomib 60 mg + Standard-of-care | Placebo + Standard-of-care
Number analyzed (Participants) | 16 | 15 | 15
Participants | 1 | 4 | 3

4. Secondary Outcome: Change in UPCR
Description: Percentage change from Baseline in Urine Protein to Creatinine Ratio (UPCR) by visit
Time Frame: Week 13, Week 25, and Week 37
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change in 24-hr UPCR value
Arm/Group | Zetomipzomib 30 mg + Standard-of-care | Zetomipzomib 60 mg + Standard-of-care | Placebo + Standard-of-care
Number analyzed (Participants) | 23 | 26 | 24
percent change in 24-hr UPCR value
  Week 13: number analyzed (Participants) | 18 | 18 | 20
  Week 13 | -33.08 (34.37) | -46.33 (55.16) | -32.27 (35.24)
  Week 25: number analyzed (Participants) | 13 | 12 | 14
  Week 25 | -37.27 (45.00) | -61.56 (50.85) | -40.33 (42.47)
  Week 37: number analyzed (Participants) | 1 | 2 | 3
  Week 37 | -68.39 (NA) — Only one participant receiving 30 mg zetomipzomib was analyzed. | -72.59 (29.91) | -23.08 (17.43)

5. Secondary Outcome: Time to Complete Renal Response and Partial Renal Response
Description: The comparison of the time to Complete Renal Response and Partial Renal Response for the zetomipzomib treatment groups (zetomipzomib 30mg and zetomipzomib 60mg) versus placebo. Hazard ratio (HR) and associated two-sided CIs are estimated using the Cox proportional hazards model. The model includes terms for treatment, the randomization stratification factors, and baseline UPCR (continuous).
Time Frame: Baseline through Week 37
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: weeks
Arm/Group | Zetomipzomib 30 mg + Standard-of-care | Zetomipzomib 60 mg + Standard-of-care | Placebo + Standard-of-care
Number analyzed (Participants) | 23 | 26 | 24
weeks
  Complete Renal Response | NA [NA to NA] — NA = Not calculable because the event of interest did not occur in a sufficient number of participants to allow estimation due to early study termination. | 26.9 [24.1 to NA] — NA = Not calculable because the event of interest did not occur in a sufficient number of participants to allow estimation due to early study termination. | NA [NA to NA] — NA = Not calculable because the event of interest did not occur in a sufficient number of participants to allow estimation due to early study termination.
  Partial Renal Response | 24.3 [12.6 to NA] — NA = Not calculable because the event of interest did not occur in a sufficient number of participants to allow estimation due to early study termination. | 12.6 [12.1 to 24.0] | 25.1 [12.4 to NA] — NA = Not calculable because the event of interest did not occur in a sufficient number of participants to allow estimation due to early study termination.
Statistical Analysis 1: Comparison: Zetomipzomib 30 mg + Standard-of-care vs Placebo + Standard-of-care; Time to complete renal response for zetomipzomib 30 mg + standard-of-care versus placebo + standard-of-care; Test type: Other — Trial was early terminated; Hazard Ratio (HR) = 0.8, 95% CI 2-sided [0.2 to 3.3]
Statistical Analysis 2: Comparison: Zetomipzomib 60 mg + Standard-of-care vs Placebo + Standard-of-care; Time to complete renal response for zetomipzomib 60 mg + standard-of-care versus placebo + standard-of-care; Test type: Other — Trial was early terminated; Hazard Ratio (HR) = 2.1, 95% CI 2-sided [0.7 to 6.7]
Statistical Analysis 3: Comparison: Zetomipzomib 30 mg + Standard-of-care vs Placebo + Standard-of-care; Time to partial renal response for zetomipzomib 30 mg + standard-of-care versus placebo + standard-of-care; Test type: Other — Trial was early terminated; Hazard Ratio (HR) = 1.3, 95% CI 2-sided [0.5 to 3.0]
Statistical Analysis 4: Comparison: Zetomipzomib 60 mg + Standard-of-care vs Placebo + Standard-of-care; Time to partial renal response zetomipzomib 60 mg + standard-of-care versus placebo + standard-of-care; Test type: Other — Trial was early terminated; Hazard Ratio (HR) = 2.6, 95% CI 2-sided [1.1 to 5.9]

6. Secondary Outcome: Proportion of Patients With UPCR ≤0.5
Description: Proportion of patients with UPCR ≤0.5
Time Frame: Week 13, Week 25, and Week 37
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Zetomipzomib 30 mg + Standard-of-care | Zetomipzomib 60 mg + Standard-of-care | Placebo + Standard-of-care
Number analyzed (Participants) | 23 | 26 | 24
Participants
  Week 13: number analyzed (Participants) | 18 | 18 | 20
  Week 13 | 2 | 5 | 2
  Week 25: number analyzed (Participants) | 13 | 12 | 14
  Week 25 | 1 | 5 | 3
  Week 37: number analyzed (Participants) | 1 | 2 | 3
  Week 37 | 0 | 1 | 0

7. Secondary Outcome: Percent Change in the Systemic Lupus Erythematosus (SLE) Disease Activity Index 2000 (SLEDAI-2K)
Description: Percent change from Baseline in clinical SLEDAI-2K score. The SLEDAI-2K score falls between 0 and 105. A higher score represents greater disease activity.
Time Frame: Week 13, Week 25, and Week 37
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change of SLEDAI-2K score
Arm/Group | Zetomipzomib 30 mg + Standard-of-care | Zetomipzomib 60 mg + Standard-of-care | Placebo + Standard-of-care
Number analyzed (Participants) | 23 | 26 | 24
percent change of SLEDAI-2K score
  Week 13: number analyzed (Participants) | 18 | 17 | 22
  Week 13 | -14.0 (45.4) | -56.4 (24.1) | -19.5 (33.7)
  Week 25: number analyzed (Participants) | 13 | 12 | 15
  Week 25 | -18.6 (45.9) | -59.2 (33.6) | -27.2 (32.6)
  Week 37: number analyzed (Participants) | 1 | 2 | 3
  Week 37 | -28.6 (NA) — Only one participant reached this timepoint. | -36.4 (51.4) | -5.0 (32.8)

8. Post Hoc Outcome: Change in UPCR
Description: Percentage change from Baseline in Urine Protein to Creatinine Ratio (UPCR) by visit
Time Frame: Week 13, Week 25, and Week 37
Population: Participants in the intent to treat set defined as the participants with Class III/IV ± Class V lupus nephritis including the participant who was actually diagnosed as Class IV and was mistakenly stratified to Pure Class V. Due to the early termination of the study, not all participants reached the timepoints for efficacy analysis and no participants completed the full 52-week treatment period.
Measure: Mean (Standard Deviation); unit: percent change in 24-hr UPCR value
Arm/Group | Zetomipzomib 30 mg + Standard-of-care | Zetomipzomib 60 mg + Standard-of-care | Placebo + Standard-of-care
Number analyzed (Participants) | 23 | 26 | 25
percent change in 24-hr UPCR value
  Week 13: number analyzed (Participants) | 18 | 18 | 21
  Week 13 | -33.08 (34.37) | -46.33 (55.16) | -34.63 (36.01)
  Week 25: number analyzed (Participants) | 13 | 12 | 14
  Week 25 | -37.27 (45.00) | -61.56 (50.85) | -40.33 (42.47)
  Week 37: number analyzed (Participants) | 1 | 2 | 3
  Week 37 | -68.39 (NA) — Only one participant receiving 30 mg zetomipzomib was analyzed. | -72.59 (29.91) | -23.08 (17.43)

9. Post Hoc Outcome: Proportion of Participants With UPCR ≤0.5
Description: Proportion of Participants With UPCR ≤0.5
Time Frame: Week 13, Week 25, and Week 37
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Zetomipzomib 30 mg + Standard-of-care | Zetomipzomib 60 mg + Standard-of-care | Placebo + Standard-of-care
Number analyzed (Participants) | 23 | 26 | 25
Participants
  Week 13: number analyzed (Participants) | 18 | 18 | 21
  Week 13 | 2 | 5 | 2
  Week 25: number analyzed (Participants) | 13 | 12 | 14
  Week 25 | 1 | 5 | 3
  Week 37: number analyzed (Participants) | 1 | 2 | 3
  Week 37 | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: Through end of study visit, up to 52 weeks
Arm/Group | Zetomipzomib 30 mg + Standard-of-care | Zetomipzomib 60 mg + Standard-of-care | Placebo + Standard-of-care
All-Cause Mortality (participants affected / at risk) | 2/27 | 1/29 | 1/28
Serious Adverse Events (participants affected / at risk) | 5/27 | 8/29 | 3/28
Other Adverse Events (participants affected / at risk) | 23/27 | 25/29 | 17/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zetomipzomib 30 mg + Standard-of-care (N=27) | Zetomipzomib 60 mg + Standard-of-care (N=29) | Placebo + Standard-of-care (N=28)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0)
Generalised oedema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Dengue fever (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis salmonella (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pseudomonas infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Injection related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Lupus vasculitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zetomipzomib 30 mg + Standard-of-care (N=27) | Zetomipzomib 60 mg + Standard-of-care (N=29) | Placebo + Standard-of-care (N=28)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (7) | 1 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 5 (10) | 5 (9) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (6) | 8 (28) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (10) | 9 (28) | 2 (2)
Asthenia (General disorders) | 0 (0) | 1 (2) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 6 (19) | 0 (0)
Face oedema (General disorders) | 0 (0) | 1 (6) | 0 (0)
Fatigue (General disorders) | 2 (3) | 0 (0) | 1 (1)
Generalised oedema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 1 (4) | 1 (1) | 1 (1)
Injection site pain (General disorders) | 0 (0) | 2 (3) | 0 (0)
Injection site reaction (General disorders) | 4 (17) | 11 (25) | 0 (0)
Injection site urticaria (General disorders) | 1 (1) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 1 (6) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 1 (1) | 1 (1)
Pain (General disorders) | 0 (0) | 2 (6) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 6 (18) | 12 (35) | 2 (3)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 3 (3) | 0 (0)
Genital herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nasal herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 4 (7) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Tinea infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 6 (6) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Blood bicarbonate decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood cholesterol increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood uric acid increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Low density lipoprotein increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Mean cell haemoglobin concentration decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 1 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (3) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (12) | 4 (10) | 2 (3)
Lethargy (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Paraparesis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Antisocial personality disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Autism spectrum disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 3 (3) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (3)
Menstruation irregular (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (5) | 1 (1)
Hypersensitivity pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Post inflammatory pigmentation change (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (5) | 2 (2)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (4) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 2 (2)
Peripheral coldness (Vascular disorders) | 0 (0) | 1 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated early for strategic business reasons following the temporary halt of the study per the Independent Data Monitoring Committee's (IDMC's) recommendation. At the time of termination, no participants had completed the full 52-week treatment period. Due to early termination, safety was the primary focus of this study and only limited efficacy data were analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-01-27): https://cdn.clinicaltrials.gov/large-docs/50/NCT05781750/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-24): https://cdn.clinicaltrials.gov/large-docs/50/NCT05781750/SAP_001.pdf